CLINICAL TRIAL: NCT04409860
Title: Randomized Controlled Trial of the Efficacy of Adjuvant Chemotherapy in Patients With Residual Lesions After Concurrent Radiochemotherapy for Locally Advanced Cervical Cancer
Brief Title: The Efficacy of Adjuvant Chemotherapy in Locally Advanced Cervical Cancer
Acronym: CQGOG0102
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Associated Director, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0102
Record Dates: First submitted 2020-05-23; First posted 2020-06-01 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Cervical Cancer
Keywords: Locally adcanced; CCRT; Adjuvant chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Observation; TP protocol; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): In this group, observation is given after CCRT.
  Interventions: Radiation: CCRT
- trial group (Experimental): In this group, adjuvant chemotherapy is given after CCRT.
  Interventions: Radiation: CCRT; Drug: Paclitaxel, Cisplatin

INTERVENTIONS:
Radiation: CCRT — Radiation concurrent platinum-containing chemotherapy (cisplatin or carboplatin)
  Other Names: control group: CCRT + observation
Drug: Paclitaxel, Cisplatin — The regimen of adjuvant chemotherapy following CCRT is Paclitaxel(150mg/m2 D1), Cisplatin(60mg/m2 D1) , q3w, three cycles.
  Other Names: trial group: CCRT + adjuvant chemotherapy
  Arms: trial group

SUMMARY:
The aim of this trial was to evaluate the efficacy of adjuvant chemotherapy in the locally advanced cervical cancer with residual lesions after concurrent chemoradiation therapy.

DETAILED DESCRIPTION:
1. Objective:

   To compare response rate and survivals of locally advanced stage cervical cancer patients with residual lesions who had CCRT alone to those who had adjuvant chemotherapy after CCRT.
2. Patients:

   1. Cervical cancer stage IIb to IVa with histopathology of squamous cell carcinoma, adenosquamous cell carcinoma, adenocarcinoma
   2. Complete CCRT(Radiation Does: A point 85Gy(+/-10%), B点50Gy(+/-10%), concurrent platinum-containing chemotherapy（cisplatin or carboplatin）
   3. MRI is performed within 4 weeks after CCRT and shows residual lesions (non-lymph node≥10mm, lymph node shortest diameter≥15mm).
3. Methods:

The patients who have residual lesions after CCRT are randomized to arm A by observation or arm B by adjuvant chemotherapy with paclitaxel plus cisplatin every 3 weeks for 3 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical cancer stage IIb to IVa with histopathology of squamous cell carcinoma, adenosquamous cell carcinoma, adenocarcinoma
2. Complete CCRT(Radiation Does: A point 85Gy(+/-10%)，B点50Gy(+/-10%)，concurrent platinum-containing chemotherapy (cisplatin or carboplatin))
3. MRI is performed within 4 weeks after CCRT and shows residual lesions (non-lymph node≥10mm, lymph node shortest diameter≥15mm).
4. ECOG<2
5. Expected survival is longer than six months
6. Hb≥70g/L、WBC≥3.5×109/ L 、ANC≥1.5×109/L、PLT≥80×109/L
7. ALT and AST≤2×ULN, Serum creatinine≤1.5×ULN
8. The serum or urine pregnancy test must be negative within 7 days before enrollment for the women of childbearing age who should agree that contraception must be used during the trial

Exclusion Criteria:

1. Activity or uncontrol severe infection
2. Liver cirrhosis, Decompensated liver disease
3. History of immune deficiency, including HIV positive or suffering from congenital immunodeficiency disease
4. Patients who cannot tolerate chemotherapy because of chronic renal insufficiency or renal failure
5. Have suffered or combined with other malignant tumor
6. Myocardial infarction, severe arrhythmia and NYHA (New York heart association)≥2 for congestive heart failure
7. A history targeted therapy or pelvic artery embolization
8. Artery-enous thrombosis within 6 months
9. Patients with autoimmune diseases
10. Complications, need to be treatment with drugs which may lead to liver or kidney injury
11. Patients with disease progression after chemoradiation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression-free survival

SECONDARY OUTCOMES:
OS | 5 years
  5 years overall survival
ORR | 3 months
  To evaluate the objective response rate(CR+PR) of adjuvant chemotherapy in cervical cancer

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Sanjose S, Serrano B, Castellsague X, Brotons M, Munoz J, Bruni L, Bosch FX. Human papillomavirus (HPV) and related cancers in the Global Alliance for Vaccines and Immunization (GAVI) countries. A WHO/ICO HPV Information Centre Report. Vaccine. 2012 Nov 20;30 Suppl 4:D1-83, vi. doi: 10.1016/S0264-410X(12)01435-1. No abstract available. PMID 23510764
- [Background] Verma J, Monk BJ, Wolfson AH. New Strategies for Multimodality Therapy in Treating Locally Advanced Cervix Cancer. Semin Radiat Oncol. 2016 Oct;26(4):344-8. doi: 10.1016/j.semradonc.2016.05.003. Epub 2016 May 26. PMID 27619255
- [Background] Rose PG. Chemoradiotherapy for cervical cancer. Eur J Cancer. 2002 Jan;38(2):270-8. doi: 10.1016/s0959-8049(01)00352-5. PMID 11803143
- [Background] Chemoradiotherapy for Cervical Cancer Meta-Analysis Collaboration. Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: a systematic review and meta-analysis of individual patient data from 18 randomized trials. J Clin Oncol. 2008 Dec 10;26(35):5802-12. doi: 10.1200/JCO.2008.16.4368. Epub 2008 Nov 10. PMID 19001332
- [Background] Chereau E, DE LA Hosseraye C, Ballester M, Monnier L, Rouzier R, Touboul E, Darai E. The role of completion surgery after concurrent radiochemotherapy in locally advanced stages IB2-IIB cervical cancer. Anticancer Res. 2013 Apr;33(4):1661-6. PMID 23564812
- [Background] Carcopino X, Houvenaeghel G, Buttarelli M, Esterni B, Tallet A, Goncalves A, Jacquemier J. Equivalent survival in patients with advanced stage IB-II and III-IVA cervical cancer treated by adjuvant surgery following chemoradiotherapy. Eur J Surg Oncol. 2008 May;34(5):569-75. doi: 10.1016/j.ejso.2007.04.006. Epub 2007 May 25. PMID 17531428
- [Background] Hequet D, Marchand E, Place V, Fourchotte V, De La Rochefordiere A, Dridi S, Coutant C, Lecuru F, Bats AS, Koskas M, Bretel JJ, Bricou A, Delpech Y, Barranger E. Evaluation and impact of residual disease in locally advanced cervical cancer after concurrent chemoradiation therapy: results of a multicenter study. Eur J Surg Oncol. 2013 Dec;39(12):1428-34. doi: 10.1016/j.ejso.2013.10.006. Epub 2013 Oct 23. PMID 24183796
- [Background] Ferrandina G, Margariti PA, Smaniotto D, Petrillo M, Salerno MG, Fagotti A, Macchia G, Morganti AG, Cellini N, Scambia G. Long-term analysis of clinical outcome and complications in locally advanced cervical cancer patients administered concomitant chemoradiation followed by radical surgery. Gynecol Oncol. 2010 Dec;119(3):404-10. doi: 10.1016/j.ygyno.2010.08.004. PMID 20817228
- [Background] Colombo PE, Bertrand MM, Gutowski M, Mourregot A, Fabbro M, Saint-Aubert B, Quenet F, Gourgou S, Kerr C, Rouanet P. Total laparoscopic radical hysterectomy for locally advanced cervical carcinoma (stages IIB, IIA and bulky stages IB) after concurrent chemoradiation therapy: surgical morbidity and oncological results. Gynecol Oncol. 2009 Sep;114(3):404-9. doi: 10.1016/j.ygyno.2009.05.043. Epub 2009 Jun 24. PMID 19555996
- [Background] Houvenaeghel G, Lelievre L, Rigouard AL, Buttarelli M, Jacquemier J, Viens P, Gonzague-Casabianca L. Residual pelvic lymph node involvement after concomitant chemoradiation for locally advanced cervical cancer. Gynecol Oncol. 2006 Jul;102(1):74-9. doi: 10.1016/j.ygyno.2005.11.037. Epub 2006 Jan 10. PMID 16406062
- [Background] Houvenaeghel G, Lelievre L, Buttarelli M, Jacquemier J, Carcopino X, Viens P, Gonzague-Casabianca L. Contribution of surgery in patients with bulky residual disease after chemoradiation for advanced cervical carcinoma. Eur J Surg Oncol. 2007 May;33(4):498-503. doi: 10.1016/j.ejso.2006.10.011. Epub 2006 Dec 6. PMID 17156969
- [Background] Vrdoljak E, Omrcen T, Novakovic ZS, Jelavic TB, Prskalo T, Hrepic D, Hamm W. Concomitant chemobrachyradiotherapy with ifosfamide and cisplatin followed by consolidation chemotherapy for women with locally advanced carcinoma of the uterine cervix--final results of a prospective phase II-study. Gynecol Oncol. 2006 Nov;103(2):494-9. doi: 10.1016/j.ygyno.2006.03.060. Epub 2006 Jun 30. PMID 16814371
- [Background] Domingo E, Lorvidhaya V, de Los Reyes R, Syortin T, Kamnerdsupaphon P, Lertbutsayanukul C, Vito-Cruz E, Tharavichitkul E, Jin K, Yoshihara M, Cupino N, Lertsanguansinchai P. Capecitabine-based chemoradiotherapy with adjuvant capecitabine for locally advanced squamous carcinoma of the uterine cervix: phase II results. Oncologist. 2009 Aug;14(8):828-34. doi: 10.1634/theoncologist.2009-0041. Epub 2009 Aug 6. PMID 19661184
- [Background] Choi CH, Lee YY, Kim MK, Kim TJ, Lee JW, Nam HR, Huh SJ, Lee JH, Bae DS, Kim BG. A matched-case comparison to explore the role of consolidation chemotherapy after concurrent chemoradiation in cervical cancer. Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1252-7. doi: 10.1016/j.ijrobp.2010.07.2006. Epub 2010 Nov 13. PMID 21075554
- [Background] Zhang MQ, Liu SP, Wang XE. Concurrent chemoradiotherapy with paclitaxel and nedaplatin followed by consolidation chemotherapy in locally advanced squamous cell carcinoma of the uterine cervix: preliminary results of a phase II study. Int J Radiat Oncol Biol Phys. 2010 Nov 1;78(3):821-7. doi: 10.1016/j.ijrobp.2009.08.069. Epub 2010 Mar 6. PMID 20207507
- [Background] Duenas-Gonzalez A, Zarba JJ, Patel F, Alcedo JC, Beslija S, Casanova L, Pattaranutaporn P, Hameed S, Blair JM, Barraclough H, Orlando M. Phase III, open-label, randomized study comparing concurrent gemcitabine plus cisplatin and radiation followed by adjuvant gemcitabine and cisplatin versus concurrent cisplatin and radiation in patients with stage IIB to IVA carcinoma of the cervix. J Clin Oncol. 2011 May 1;29(13):1678-85. doi: 10.1200/JCO.2009.25.9663. Epub 2011 Mar 28. PMID 21444871
- [Background] Tang J, Tang Y, Yang J, Huang S. Chemoradiation and adjuvant chemotherapy in advanced cervical adenocarcinoma. Gynecol Oncol. 2012 May;125(2):297-302. doi: 10.1016/j.ygyno.2012.01.033. Epub 2012 Jan 31. PMID 22307061
- [Background] Lorvidhaya V, Chitapanarux I, Sangruchi S, Lertsanguansinchai P, Kongthanarat Y, Tangkaratt S, Visetsiri E. Concurrent mitomycin C, 5-fluorouracil, and radiotherapy in the treatment of locally advanced carcinoma of the cervix: a randomized trial. Int J Radiat Oncol Biol Phys. 2003 Apr 1;55(5):1226-32. doi: 10.1016/s0360-3016(02)04405-x. PMID 12654431
- [Background] Tangjitgamol S, Tharavichitkul E, Tovanabutra C, Rongsriyam K, Asakij T, Paengchit K, Sukhaboon J, Penpattanagul S, Kridakara A, Hanprasertpong J, Chomprasert K, Wanglikitkoon S, Atjimakul T, Pariyawateekul P, Katanyoo K, Tanprasert P, Janweerachai W, Sangthawan D, Khunnarong J, Chottetanaprasith T, Supawattanabodee B, Lertsanguansinchai P, Srisomboon J, Isaranuwatchai W, Lorvidhaya V. A randomized controlled trial comparing concurrent chemoradiation versus concurrent chemoradiation followed by adjuvant chemotherapy in locally advanced cervical cancer patients: ACTLACC trial. J Gynecol Oncol. 2019 Jul;30(4):e82. doi: 10.3802/jgo.2019.30.e82. Epub 2019 Apr 10. PMID 31074236